CLINICAL TRIAL: NCT00214435
Title: A Randomised, Multi-Centre, Open-Label Study in Well-Controlled Treatment-Experienced HIV-Infected Patients to Assess Compliance With a Once-Daily Regimen of Lamivudine, Efavirenz and Didanosine Versus Continuation of Current Anti-Retroviral Regimen Delivered at Least Twice Daily
Brief Title: Once Daily 3TC, Efavirenz and ddI for HIV Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 407 Doctors (Other)
Collaborators: Bristol-Myers Squibb (Industry); Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TEddI
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infection; AIDS
Keywords: HIV infection; AIDS; Adherence; MEMS caps; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Drug: once daily minimum 3-drug regimen of anti-retroviral medications

SUMMARY:
Poor compliance is thought to be a major cause of treatment failure. The TEddI study is a randomised, multi-centre, open-label study in well-controlled treatment-experienced HIV-infected patients to assess compliance with a once-daily regimen of antiretroviral therapy versus continuation of current anti-retroviral regimen delivered at least twice daily.

DETAILED DESCRIPTION:
Rationale: 'TEddI' will enable a once-daily treatment strategy to be studied and provide information on effectiveness, patient adherence and quality of life and the tolerability of such regimens.

Hypothesis: The study hypothesis is that an antiretroviral regimen comprising of three agents taken once daily will have higher levels of adherence than a regimen requiring more frequent dosing.

Primary objective: To determine over 24 weeks the levels of adherence in two groups of HIV-infected subjects randomised to receive either a once daily minimum 3-drug regimen or to continue a minimum 3-drug regimen requiring more frequent dosing.

Secondary objectives: The secondary objectives of the study will include:

* To estimate the proportion of patients with treatment failure where treatment failure is defined as:
* HIV-1 RNA viral load of >400 copies/ml on two consecutive occasions more than one month apart, OR
* Discontinuation of treatment for any reason (where subsequent therapy does not comply with the study regimen change guidelines outlined in section 3.3.3)
* Proportion of patients with plasma HIV-RNA less than 50 copies/ml (using an ultrasensitive assay) at 24 and 48 weeks
* Change from baseline in CD4 cell count at 24 and 48 weeks
* Changes from baseline in subjects' quality of life at 24 and 48 weeks
* Changes from baseline based on DASS 21 scores at 24 and 48 weeks
* Incidence and severity of adverse events and abnormal laboratory values (grade 3 & 4) at 24 and 48 weeks
* Proportion of patients remaining on assigned treatment Study Design This is a randomised, open-label, multi-centre, prospective, 48-week study comparing a 3 (or more) drug once-daily antiretroviral regimen with any 3 (or more) drug regimen in which at least 1 drug must be taken at least twice daily.

One hundred and twenty (120) subjects will be recruited and randomised in a 1:1 ratio to one of two open-label treatment regimens and will continue to receive randomised treatment until week 24:

Arm 1: (Once daily arm) commence treatment with a once-a-day combination of licensed antiviral medications (such as EFV/ddI/3TC, EFV/3TC/TDF or ATV/3TC/TDF).

Arm 2: (Continuation arm) continue current ART (minimum 3-drugs) dosed twice daily or more frequently

Following week 24, patients will have the option to continue randomised treatment for a further 24 weeks or switch to the once daily treatment arm. In all cases, patients will be followed up for 48 weeks from the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or more with laboratory evidence of HIV-1 infection
* ability to understand and provide written informed consent to participate in the study
* stable on current ART regimen for at least 3 months prior to screening.
* plasma HIV-RNA less than 400 copies/ml at the screening visit.
* women of child bearing potential must have a negative serum or urine β-HCG pregnancy test within 14 days prior to week -4 (assessment of study eligibility)

Exclusion Criteria:

* virological failure of a proposed Once daily arm medication
* a serious medical condition which may compromise the subject's safety, including an active AIDS-defining condition within the previous 6 months
* known toxicities to any of the proposed Once daily arm medications
* laboratory abnormalities at screening:
* serum creatinine greater than twice the upper limit of normal (2 x upper limit of normal (ULN))
* AST, ALT or alkaline phosphatase greater than 5 times the ULN
* lactate greater than 2.5 x ULN
* haemoglobin less than 9.5 g/dL
* women who are pregnant or breast-feeding or who, if of child-bearing potential, are not willing to use adequate contraception (including barrier contraception)
* patients who in the investigator's opinion are unlikely to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-05

PRIMARY OUTCOMES:
- levels of adherence

SECONDARY OUTCOMES:
- proportion of patients with treatment failure where treatment failure is defined
- HIV-1 RNA viral load of >400 copies/ml on two consecutive occasions more than one month apart, OR discontinuation of treatment for any reason (where subsequent therapy does not comply with the study regimen change guidelines outlined in section 3.3.3)
- proportion of patients with plasma HIV-RNA less than 50 copies/ml (using an ultrasensitive assay) at 24 and 48 weeks
- change from baseline in CD4 cell count at 24 and 48 weeks
- changes from baseline in subjects' quality of life at 24 and 48 weeks
- changes from baseline based on DASS 21 scores at 24 and 48 weeks
- incidence and severity of adverse events and abnormal
- laboratory values (grade 3 & 4) at 24 and 48 weeks
- proportion of patients remaining on assigned treatment

CONTACTS AND LOCATIONS:
Overall Officials: David A Baker, MB ChB, Principal Investigator — 407 Doctors
Locations (1):
- 407 Doctors, Sydney, New South Wales, Australia